CLINICAL TRIAL: NCT04280640
Title: LCCC 1938: Investigating the Relationship Between Circulating Tumor Cell Cultures Treatment Response and Clinical Outcomes
Brief Title: Relationship Between Circulating Tumor Cell Cultures' Treatment Response and Clinical Outcomes
Status: Withdrawn | Type: Observational
Why Stopped: PI left UNC.
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC1938
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Cancer; Metastasis Lung; Metastasis to Liver; Circulating Tumor Cell; Gastrointestinal Cancer; Bladder Cancer
MeSH Terms: conditions — Neoplasms; Neoplastic Cells, Circulating; Gastrointestinal Neoplasms; Urinary Bladder Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Metastatic Cancer Pts Receiving Molecularly Targeted Therapy: Metastatic cancer patients (with liver and/or lung metastasis) who will receive molecularly targeted therapy based on genomic testing data
  Interventions: Other: Blood Draw
- GI Cancer Pts: Gastrointestinal cancer patients (with liver and/or lung metastasis) who will receive 3rd line treatments or enrolled on a targeted therapy treatment trial
  Interventions: Other: Blood Draw
- Bladder Cancer Pts: Bladder cancer patients (with liver and/or lung metastasis) who will receive systemic treatment
  Interventions: Other: Blood Draw

INTERVENTIONS:
Other: Blood Draw — A blood sample will be collected once, prior to treatment.

SUMMARY:
The purpose of this prospective, non-randomized, single-center pilot exploratory study is to investigate whether established circulating tumor cell (CTC) cultures have a similar response to targeted therapy treatment as the in vivo (patients') disease.

DETAILED DESCRIPTION:
This study will isolate circulating tumor cells (CTCs) from blood samples taken from patients with liver and/or lung metastases who will receive systemic treatments. The CTCs will be cultured and given the same treatment as the patient received. The main goals of this project are 1) to assess CTC cultures' treatment response and compare the in vitro response to the clinical response, and 2) determine the sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) of CTC cultures' response in predicting clinical response including complete response (CR), partial response (PR), stable disease (SD) and progressive disease (PD).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a metastatic solid tumor malignancy with either liver and/or lung metastasis. Patients with newly diagnosed metastatic disease who have not had systemic therapy or are progressing on systemic therapy fitting one of the following cohorts:

  * Patients had a tumor or liquid biopsy with molecular analysis (genomic analysis or other type of molecular characterization) resulting in a therapeutic target with planned targeted therapy by the patient's treating physician.
  * Gastric cancer patients who have failed the first and second line chemotherapy.
  * Bladder cancer patients (with liver and/or lung metastasis) who will receive systemic treatment.
* Scheduled to initiate systemic treatment for management of their disease. The systemic treatment will be either cytotoxic chemotherapy or targeted therapy but not checkpoint inhibitor immunotherapy.
* ≥18 years of age
* Written informed consent obtained and signed
* Able to have blood collection without excessive difficulty

Exclusion Criteria:

* Patient unwilling or unable to complete informed consent
* Currently pregnant or lactating women
* Physical or psychological inability to complete sample collection for any reason including but not limited to: inability to tolerate any study procedures, any physical limitation that would undermine the safety of the subject in the study, or any psychiatric or neurological condition that inhibits full comprehension of study requirements and inability to complete informed consent, as determined by treating physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients with liver and/or lung metastasis who will receive systemic treatment.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Correlation between treatment response in CTCs and in vivo | Initiation of trial to 24 months post-initiation
  To estimate the agreement between CTC cultures' response to treatment, dichotomized as either yes or no response, to the clinical response in patients to treatment, dichotomized as either progressive disease (PD) versus complete response (CR), partial response (PR), or stable disease (SD)

SECONDARY OUTCOMES:
Sensitivity, specificity, and predictive values of CTC cultures' treatment response | Initiation of trial to 24 months post-initiation
  To determine the sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) of CTC cultures' response in predicting clinical response including complete response (CR), partial response (PR), stable disease (SD) and progressive disease (PD)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Z Wang, MD, Principal Investigator — UNC Chapel Hill